CLINICAL TRIAL: NCT03172572
Title: Outcomes After Minimally Invasive or Open Pancreatoduodenectomy in High-volume Centers; a Pan-European Retrospective Propensity-score Matched Cohort Study
Brief Title: A Pan-European Study on Minimally Invasive Versus Open Pancreatoduodenectomy in High-volume Centers
Acronym: MI-PD
Status: Completed | Type: Observational
Sponsor: S (Sjors) Klompmaker, MD (Other)
Responsible Party: Sponsor-Investigator, S (Sjors) Klompmaker, MD, PhD Candidate, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: W16_401#17.011
Record Dates: First submitted 2017-05-26; First posted 2017-06-01 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Pancreatic Neoplasms; Pancreas Cyst; Pancreas Cancer
Keywords: minimally invasive surgical procedures; pancreas surgery; pancreatoduodenectomy
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Indication for surgery: Solid neoplasms
  Interventions: Procedure: Minimally invasive pancreatoduodenectomy; Procedure: Open pancreatoduodenectomy

INTERVENTIONS:
Procedure: Minimally invasive pancreatoduodenectomy — Laparoscopic, robot-assisted, or hybrid resection
Procedure: Open pancreatoduodenectomy — Open resection

SUMMARY:
RATIONALE: Minimally-invasive pancreatoduodenectomy (MIPD), either laparoscopic or robot-assisted, has been suggested as a valuable alternative to open pancreatoduodenectomy (OPD). The generalizability of the current literature is, however, unknown since randomized studies are lacking, and current data are published from few, very high volume centers and selection bias with a lack of case-matched series. International studies are lacking completely.

OBJECTIVE: To compare outcomes of MIPD versus open pancreatoduodenectomy (OPD), in high-volume European pancreas centers (>10 MIPDs per year, total >20 PDs per year).

METHODS: A retrospective multicenter propensity-score matched cohort study including all consecutive patients who underwent MIPD (or MI total pancreatectomy) between January 2012 and December 2016, for pancreatic head, bile duct, or duodenal cancer or cysts except chronic pancreatitis. Predefined electronic case report forms will be disseminated amongst participating centers. Participants are responsible for their own data collection. Matching of MIPD cases (collected from participating centers) to OPD controls (extracted from Dutch and German national registries) will be based on propensity scores determined by logistic regression including preoperative variables: year of surgery, demographics, BMI, ASA, comorbidities, tumor size, tumor etiology (diagnosis), and multivisceral resection. Primary outcome is 90-day major morbidity(Clavien-Dindo ≥ 3a). Secondary outcomes are 90-day postoperative events including: pancreatic fistula, length of hospital stay, R0 (microscopically negative) resection margin, malignant lymph node ratio, days to adjuvant therapy and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Indication for open or minimally invasive pancreatoduodenectomy
* Pancreatic head, bile duct, or duodenal cancer or cysts

Exclusion Criteria:

* Chronic pancreatitis without suspected solid tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases (minimally-invasive pancreatoduodenectomy) will be retrieved from participating high-volume centers (2012 and 2017).
  Controls (open pancreatoduodenectomy) will be retrieved from German and Dutch population-based pancreatic surgery registries (2015-2017).
Sampling Method: Non-Probability Sample
Enrollment: 4220 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Major morbidity | 90-days
  Clavien-Dindo grade 3a-5 complications

SECONDARY OUTCOMES:
Pancreatic fistulae | 90-days
  ISGPS 2017 definition
Length of stay | 90-days
  length of hospital stay
Radical resection rate | 90-days
  R0/R1/R2 classification
Malignant lymph node ratio | 90-days
  Malignant/ non-malignant lymph nodes
time to adjuvant therapy | 90-days
  Resection to adjuvant chemo(-radio) therapy
Overall survival | 90-days

CONTACTS AND LOCATIONS:
Locations (1):
- Sjors Klompmaker, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klompmaker S, van Hilst J, Wellner UF, Busch OR, Coratti A, D'Hondt M, Dokmak S, Festen S, Kerem M, Khatkov I, Lips DJ, Lombardo C, Luyer M, Manzoni A, Molenaar IQ, Rosso E, Saint-Marc O, Vansteenkiste F, Wittel UA, Bonsing B, Groot Koerkamp B, Abu Hilal M, Fuks D, Poves I, Keck T, Boggi U, Besselink MG; European consortium on Minimally Invasive Pancreatic Surgery (E-MIPS). Outcomes After Minimally-invasive Versus Open Pancreatoduodenectomy: A Pan-European Propensity Score Matched Study. Ann Surg. 2020 Feb;271(2):356-363. doi: 10.1097/SLA.0000000000002850. PMID 29864089
- See also: Consortium Website — http://www.e-mips.org/mipd/